CLINICAL TRIAL: NCT05518617
Title: Molecular and Functional Imaging of Parkinson's Pathology in SNCA, Parkin and PINK1 Mutation Carriers
Brief Title: Molecular and Functional Imaging in Monogenic PD.
Acronym: FOX_1
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-21-14
Record Dates: First submitted 2022-07-25; First posted 2022-08-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Nervous System Disorder; Neurodegenerative Diseases; Neurodegenerative Disease, Hereditary; Parkinson's
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases; Neurodegenerative Diseases; Heredodegenerative Disorders, Nervous System | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biosamples collected during this study will be blood, urine, and CSF. Blood biomarkers include routine clinical laboratory, DNA testing, and other analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- SNCA (Alpha-synuclein gene): PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology.
  Interventions: Other: Positron Emission Tomography (PET) scan using DASB tracer
- Parkin (Parkin gene): PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology
  Interventions: Other: Positron Emission Tomography (PET) scan using DASB tracer
- PINK1 (Phosphatase and Tensin Homolog (PTEN)-Induced Kinase 1 gene): PET and SPECT molecular imaging and MRI; Clinical investigation and computerized neuropsychological testing; Collection of blood, urine and CSF biomarkers of PD pathology
  Interventions: Other: Positron Emission Tomography (PET) scan using DASB tracer
- GBA1 (Glucosylceramidase beta gene): Symptomatic and asymptomatic heterozygous carriers of risk variants to the GBA1 gene for Parkinson's disease

INTERVENTIONS:
Other: Positron Emission Tomography (PET) scan using DASB tracer — DASB is a highly selective PET radioligand for serotonin transporter and is a reliable tool to investigate serotonin terminals and neurons.
  The included Magnetic Resonance Imaging (MRI) sequences serve to provide additional information plus complement PET data.
  To quantify dopaminergic pathology with [123I]FP-CIT SPECT,
  Other Names: FP-CIT Single-photon Emission Computed Tomography (SPECT) scan; Magnetic Resonance Imaging (MRI) Scan; Lumbar puncture
  Groups: PINK1 (Phosphatase and Tensin Homolog (PTEN)-Induced Kinase 1 gene); Parkin (Parkin gene); SNCA (Alpha-synuclein gene)

SUMMARY:
In this study, the investigators aim to find a biomarker of Parkinson's disease. This is done using imaging scans called Positron Emission tomography (PET), Single Photon Emission Computed Tomography (SPECT), and Magnetic Resonance Imaging (MRI). The findings will provide a deeper understanding of the brain changes in Parkinson's disease. More importantly, this study will help with the discovery and development of new medications aiming to delay progression of PD symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to find a biomarker for Parkinson's disease (PD). A biomarker is an indicator of the presence of a disease, that can be measured, and that is able to give information about the progression, or severity, of it.

PD is a chronic neurological disease that progresses over time and causes a variety of symptoms, such as slowness of movement, stiffness and shaking. The symptoms of PD are caused by the malfunction and death of vital nerve cells in the brain. it is no known what causes PD and there is no biomarker for it.

Generally, PD occurs without a known cause, and is called sporadic PD. In a few cases, however, PD occurs because of a genetic mutation, and it is called genetic PD. Patients with genetic PD share features to sporadic PD patients. It is believed that studying people who carry mutations for genetic PD mutations would provide precious information on what are the causes of PD and help to devise successful treatments.

Participants will attend 4 visits in a 3 month period. These visits include an initial consent and assessment visit where some blood samples will also be taken. the second visit involves a PET scan with the tracer DASB along with an MRI scan. The third visit involves a SPECT scan. the fourth visit is optional and would be for a lumbar puncture visit. Each visit will last around 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be judged by the investigator able to understand the nature, design, and procedures of the study and must be able to provide a signed and dated informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* All subjects must be willing and able to comply with scheduled visits, required study procedures and laboratory tests.
* All subjects must be able to travel to the research sites for the study procedures.
* For female subjects: They must be either of non-childbearing potential (either surgically sterile or post- menopausal - defined as 12 months of spontaneous amenorrhea), or, if of childbearing potential, subjects must demonstrate to be non-pregnant (as demonstrated by negative urine β-HCG test at screening), non-breastfeeding.
* All subjects must comply with highly effective contraceptive measures. A highly effective contraceptive measure is defined as a measure that can achieve a failure rate of less than 1% per year when used consistently and correctly. These methods are listed in more detail below:

Oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation;

Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation:

Intrauterine device (IUD)

Intrauterine hormone-releasing system (IUS)

Bilateral tubal occlusion

Vasectomised partner

Sexual abstinence

* For sexually active male subjects, they must agree to use condoms to protect their partners from becoming pregnant for the duration of the study and for 3 months after the last administration of PET or SPECT ligands. They must also agree to ensure that they and their partners are routinely using a medically approved contraceptive method. It is important that male subjects not impregnate others for the duration of the study and for 3 months after the last administration of PET or SPECT ligands.

  **All subjects must have adequate visual and auditory acuity according to investigator's judgement to complete the psychological testing.
* All subjects must have no use of medications with known interaction with serotonergic transmission (e.g. selective serotonin reuptake inhibitors, tricyclic antidepressant, triptans, etc).
* For subjects taking any drugs that might interfere with dopamine transporter SPECT imaging (neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative) must be willing and able from a medical standpoint to hold the medication for at least 5 half-lives prior to screening DaTSCANä imaging.

Exclusion Criteria:

* Subjects lacking capacity according to investigator judgement.
* Subjects with a clinical diagnosis of dementia as determined by the investigator.
* Current treatment with anticoagulants (e.g. warfarin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Use of any of the following drugs that might interfere with dopamine transporter SPECT imaging: neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 5 months of Screening.
* Use of investigational drugs or devices within 60 days prior to Baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).
* History of cancer within the last 5 years, with the exception of non-metastatic basal cell carcinoma of the skin.
* Subjects with current or recent history of drug or alcohol abuse/dependence.
* Contraindication to MRI, such as presence of metal devises or implants (e.g. pacemaker, vascular- or heart- valves, stents, clips), metal deposited in the body (e.g. bullets or shells), or metal grains in the eyes;
* Claustrophobia or history of back pain that makes prolonged laying on the PET or MRI scanner intolerable.
* Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort of asymptomatic and symptomatic carriers of genetic mutations for familial forms of Parkinson's Disease, and previously collected data from healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
DASB (a marker of Serotonin transporter) used to quantify in vivo pathology of serotonin | 3 weeks
  To quantify serotonergic pathology with [11C]3-amino-4-(2- imethylaminomethylphenylsulfanyl)-benzonitrile (DASB) Positron Emission Tomography (PET)
SPECT to measure brain molecular pathology | 3 weeks
  To quantify serotonergic pathology with [11C]DASB PET and dopaminergic pathology with Single-photon Emission Computed Tomography (SPECT)
Magnetic Resonance Imaging (MRI) | 3 weeks
  Magnetic Resonance Imaging (MRI) to view structural and microstructural changes and structural connectivity.

OTHER OUTCOMES:
Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) to determine if there is a correlation with neuropsychological and behavioural evaluation. | 3 weeks
  A rating tool used to gauge the course of Parkinson's disease in patients
Montreal Cognitive Assessment (MOCA) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 weeks
  A cognitive screening test designed to assist in the detection of mild cognitive impairment. Scored out of 30.
Cambridge Neuropsychological Test Automated Battery (CANTAB) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  Administered to detect cognitive issues & brain disorders efficiently.
Symbol Digit Modalities Test (SDMT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  To be used in screening for organic cerebral dysfunction sored out of 110
Beck Depression Inventory-II (BDI-II) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  A brief, self-report inventory designed to measure the severity of depression symptomatology
State-Trait Anxiety Inventory (STAI) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  A commonly used measure of trait and state anxiety. Used to diagnose anxiety and to distinguish it from depressive syndromes
University of Pennsylvania Smell Identification Test to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 Weeks
  This is used to test the function of an individual's olfactory system
Movement Disorder Society- Non-Motor Symptoms scale for Parkinson's Disease MDS-NMSS to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 weeks
  This is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease
Scales for Outcomes in Parkinson's Disease-Autonomic questionnaire - Autonomic Dysfunction (SCOPA-AUT) to determine if there is a correlation with neuropsychological and behavioural evaluation | 3 weeks
  A 25 item assessment to evaluate autonomic symptoms in patients with Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Marios Politits, Professor, Principal Investigator — The University of Exeter
Locations (1):
- University Of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Yet to be confirmed.

REFERENCES:
- See also: University of Exeter, Project infromation — https://medicine.exeter.ac.uk/clinical-biomedical/research/nig/currentstudies/